CLINICAL TRIAL: NCT00844233
Title: A Single Arm Phase II Study of Neoadjuvant Therapy Using Irinotecan Bead in Patients With Resectable Liver Metastases From Colorectal Cancer
Brief Title: Study of Chemoembolisation Using Irinotecan Bead Prior to Surgery in Metastatic Colorectal Cancer
Acronym: PARAGON-II
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA1016
Record Dates: First submitted 2009-02-09; First posted 2009-02-16 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Irinotecan Bead
  Interventions: Device: Irinotecan Bead

INTERVENTIONS:
Device: Irinotecan Bead — Irinotecan eluting bead
  Other Names: Irinotecan Bead, PARAGON Bead

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of Irinotecan Bead in the neoadjuvant treatment (i.e. the Irinotecan Bead is administered prior to surgery) of resectable liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
The Primary Endpoint of this study is Tumour resectability at surgery. Secondary Endpoints:

1. Safety assessed by SAE and AE monitoring (NCI CTCAE v3.0)
2. Tumour response assessed by imaging (RECIST and necrosis)
3. Viable residual tumour assessed by pathological evaluation of resected liver tissue.
4. Recurrence (time and site) following resection
5. Correlation of tumour response by imaging and pathology

ELIGIBILITY:
Inclusion criteria

1. Presence of potentially resectable colorectal cancer liver metastases, with less than 60% liver tumour replacement. The consulting surgeon, according to local practice, will determine resectability.
2. Patients having undergone complete resection of the primary tumour without gross or microscopic evidence of residual disease (R0), or the primary tumour is considered R0 resectable at screening.
3. Age: 18-80 years.
4. ECOG Status ≤2.
5. No previous irinotecan-containing chemotherapy for advanced disease.
6. Previous chemotherapy is allowed (unless it contained irinotecan), but must have ended at least one month prior to study entry.
7. Presence of adequate contraception in fertile (M/F) patients. Pregnant or lactating women are excluded.
8. Absence of any other previous malignancy other than adequately treated in situ carcinoma of the cervix or non-melanoma skin cancer (unless there has been a disease-free interval of at least 10 years).
9. Patients should not have participated in another clinical trial with any investigational drug in the 30 days prior to enrolment.
10. Absence of:

    * Peripheral neuropathy (CTC > grade 1)
    * Uncontrolled congestive heart failure or angina pectoris, or hypertension or arrhythmia.
    * History of significant neurologic or psychiatric disorders
    * Active infection
11. Written informed consent according to ICH/EU GCP, and any applicable local, national or international regulations.
12. Patients with liver-dominant disease, defined as ≥80% of the tumour body burden confined to the liver. Unilobar disease, or bilobar disease suitable for treatment in a single chemoembolisation procedure, with a maximum of 4 lesions.
13. Hematologic function: WBC ≥3.0 x 10*9/L, platelets ≥100 x 10*9/L, Absolute neutrophil count > 1.5 x 10*9/l.
14. Adequate organ function as measured by:

    1. Serum creatinine ≤2 x upper limit of normal (ULN).
    2. Serum transaminases (AST & ALT) ≤5 x ULN.
    3. Total bilirubin ≤1.5 x ULN.
    4. Prothrombin time >50% of normal.

Exclusion criteria

1. Extrahepatic metastases constituting >20% of tumour body burden.
2. Contraindications to irinotecan:

   1. Chronic inflammatory bowel disease and/or bowel obstruction.
   2. History of severe hypersensitivity reactions to irinotecan hydrochloride trihydrate.
   3. Severe bone marrow failure.
   4. Concomitant use with St John's Wort.
3. Active bacterial, viral or fungal infection within 72 hours of study entry.
4. Allergy to contrast media that cannot be managed with standard care.
5. Any contraindication for hepatic embolisation procedures:

   1. porto-systemic shunt.
   2. hepatofugal blood flow.
   3. severe atheromatosis.
6. Contraindication to hepatic artery catheterisation, such as a patient with severe peripheral vascular disease precluding catheterisation.
7. Other significant medical or surgical condition, or any medication or treatment regimens, that would place the patient at undue risk, that would preclude the safe use of chemoembolisation or would interfere with study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2011-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Tumour resectability at surgery | 1 month

SECONDARY OUTCOMES:
Safety assessed by SAE and AE monitoring (NCI CTCAE v3.0) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Professor Graeme Poston, MB, MS, FRCS, Principal Investigator — Consultant General Surgeon
Locations (5):
- Medical University Vienna, AKH, Vienna, Austria
- Centre Hépato-Biliaire, Hôpital Paul Brousse, Villejuif, France
- United Kingdom (3):
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke
  - University Hospital Aintree, Liverpool
  - North Manchester General Hospital, Manchester

REFERENCES:
- [Derived] Jones RP, Malik HZ, Fenwick SW, Terlizzo M, O'Grady E, Stremitzer S, Gruenberger T, Rees M, Plant G, Figueras J, Albiol M, Adam R, Awad S, Poston GJ. PARAGON II - A single arm multicentre phase II study of neoadjuvant therapy using irinotecan bead in patients with resectable liver metastases from colorectal cancer. Eur J Surg Oncol. 2016 Dec;42(12):1866-1872. doi: 10.1016/j.ejso.2016.07.142. Epub 2016 Aug 10. PMID 27561844
- [Derived] Jones RP, Dunne D, Sutton P, Malik HZ, Fenwick SW, Terlizzo M, O'Grady E, Koelblinger C, Stattner S, Stremitzer S, Gruenberger T, Poston GJ. Segmental and lobar administration of drug-eluting beads delivering irinotecan leads to tumour destruction: a case-control series. HPB (Oxford). 2013 Jan;15(1):71-7. doi: 10.1111/j.1477-2574.2012.00587.x. Epub 2012 Oct 16. PMID 23216781
- See also: Sponsor company website — http://www.biocompatibles.com